CLINICAL TRIAL: NCT00774176
Title: Pennsylvania Study of Chronic Obstructive Pulmonary Exacerbations (PA-SCOPE)
Brief Title: Pennsylvania Study Of Chronic Obstructive Pulmonary Exacerbations
Acronym: PA-SCOPE
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: PA DOH RFA-02-07-20
Record Dates: First submitted 2008-01-04; First posted 2008-10-17 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; COPD Exacerbation; Genetic markers COPD; Gene expression in COPD exacerbations; COPD Exacerbation Symptom Reporting; COPD Exacerbation Disease Management; COPD Treatment; Breathing disorders; Emphysema; COPD with Healthy Control comparators for genetic association studies.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Emphysema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Ancillary studies collect blood specimens for gene expression and genetic factors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Phase 1 & Gene Expression:Hospitalized COPD exacerbators
- 2: Phase 2: COPD group
- 3: Genetic Association Studies: COPD and Healthy Controls

SUMMARY:
The overall purpose of PA-SCOPE is to determine why black and rural residents of Pennsylvania might be at higher risk for deadly, debilitating, and costly hospitalizations for chronic obstructive pulmonary disease (COPD)- and then to show that repeat acute exacerbations in high-risk patients can be reduced with one simple intervention. We believe that 1) COPD patients who are black or who live in rural areas of Pennsylvania are at higher risk of acute exacerbations requiring hospitalization and 2) this elevated risk can be reduced with one simple intervention: access to a 1-800 Temple Call Center where patients can get immediate customized advice on managing COPD exacerbations in their early stages. We will test these beliefs in PA-SCOPE. The collaborators with Temple University Hospital on the PA-SCOPE project are Lancaster General Hospital, Western Pennsylvania Hospital, and the Philadelphia College of Osteopathic Medicine.

DETAILED DESCRIPTION:
* Overall objective: To determine why African American and rural residents of Pennsylvania might be at higher risk for deadly, debilitating, and costly hospitalizations for COPD-and to show that repeat acute exacerbations in high-risk patients can be reduced with one simple intervention--access to a 1-800 Temple Call Center phone number where patients can get immediate customized advice on managing COPD exacerbations in their early stages.
* Phase 1: To compare and contrast the influence of race and geographic location in COPD exacerbation in relation to severity, comorbidities, treatment patterns, infection rate. To identify potential risk factors for COPD exacerbations leading to hospitalization.
* Phase 2: To reduce hospitalizations and deaths due to COPD exacerbations and to improve patient quality of life, lung function, and everyday activity levels

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 & Gene Expression: --Current hospitalization for COPD exacerbation
* Phase 1 & 2: COPD & ONE of the following criteria:

  1. History of hospitalization for COPD exacerbation, OR
  2. Currently on supplemental oxygen, OR
  3. History of evaluation for lung transplant or LVRS, OR
  4. >/= 6 months post-LVRS
* Phase 1 or 2:

  1. Current or former smoker, >/= 20 pack-yr. smoking history
  2. FEV1 </= 70%; FEV1/FVC </= 70%
  3. Life expectancy of > 6 months

Exclusion Criteria:

* < 20 pack-yr. smoking history
* Diagnosis of pulmonary fibrosis, bronchiectasis, mediastinal mass, or presence of a pulmonary mass
* Asthma
* FEV1 > 70% or FEV1/FVC >70%

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Phase 1: inpatients hospitalized for COPD exacerbations Phase 2: Moderate to severe COPD
Sampling Method: Non-Probability Sample
Enrollment: 1066 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Phase 1 identifies the demographic & genetic factors affecting inpatient hospitalization for COPD exacerbation.Phase 2 documents the number of physician & ER visits, hospitalizations & death related to exacerbations. | Phase 1 is up to 10 weeks. Phase 2 is up to 2 years.

SECONDARY OUTCOMES:
Phase 2 also documents the number, severity, & subject reporting of exacerbations, spirometry changes,& quality of life. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerard J Criner, MD, Principal Investigator — Temple University
Locations (3):
- United States (3):
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Busch R, Qiu W, Lasky-Su J, Morrow J, Criner G, DeMeo D. Differential DNA methylation marks and gene comethylation of COPD in African-Americans with COPD exacerbations. Respir Res. 2016 Nov 5;17(1):143. doi: 10.1186/s12931-016-0459-8. PMID 27814717
- See also: Publication of results: PMID: 26259074 — https://www.ncbi.nlm.nih.gov/pubmed/26259074